CLINICAL TRIAL: NCT01647919
Title: Effects of cogniVida™ on Learning and Memory and in Comparison to Placebo After Long-term Supplementation
Acronym: MemIprov
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2012-01-10-STEV
Record Dates: First submitted 2012-06-22; First posted 2012-07-24 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Cognition; Attention; Memory; Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cogniVida™ 100 mg/day (Experimental)
  Interventions: Dietary Supplement: cogniVida™ 100 mg/day
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cogniVida™ 100 mg/day — 4 capsules 25 mg (total 100 mg) cogniVida™ once a day
  Arms: cogniVida™ 100 mg/day
Dietary Supplement: Placebo — 4 capsules of placebo identical to cogniVida™ once a day
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the efficacy of cogniVida™ on learning and memory performance (executive function, associative, spatial and verbal memory) as well as on mood and attention parameters after four, eight and eleven weeks of supplementation and in comparison with placebo.

cogniVida™ is considered a dietary supplement, and therefore it is not an approved drug by the Food and Drug Administration (FDA). It is regulated like a food. The U.S. Food and Drug Administration does not strictly regulate herbs and dietary supplements. The investigators do not claim that this supplement is meant to treat any ailment.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females, age 50 - 65 years
* Subject agrees to maintain his or her habitual diet and physical activity patterns throughout the study period.
* Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
* Subject has a body mass index (BMI) of ≥18.5 and ≤ 30.00 kg/m2 at screening.
* Subject is willing to refrain from consuming alcoholic drinks 24 h prior to test days and until the end of each assessment period and refrain from consuming caffeine, and caffeine-containing products 12 h prior to test days and until the end of each assessment period.
* Subject is willing to refrain from vigorous physical activity 12 h prior to test days.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subject has a positive drug screening of amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, 3,4-methylenedioxymethamphetamine, opiates or tricyclic antidepressants at screening or at any of the admission days.
* Subjects has a positive breath alcohol and breath carbon monoxide test at screening or at any of the admission days.
* Subject has abnormal clinical chemistry and hematology laboratory test results of clinical significance according to established criteria.
* Subjects with a history of renal or hepatic disease that is likely to interfere with the metabolism or excretion of the test product.
* Subject has donated more than 300 mL of blood during the three months prior to screening.
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the average blood pressure measured at screening.
* Subject has a history, in the judgment of the Investigator, of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Excessive habitual caffeine consumption (>500 mg caffeine/d), following screening and throughout the study period. Caffeine consumption will be assessed using the Caffeine Consumption Questionnaire
* Subjects who are on a significant hypocaloric diet (i.e. < 1200 calories per day) aiming for significant weight loss.
* Use of any sleep aid medication within four days prior to each test day (visits 2, 3, 4, 5; days 0, 28, 56, 77).
* Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Subject is pregnant, planning to be pregnant during the study period, lactating, or women who consider themselves to be of childbearing potential and who are engaged in an active sex life who are unwilling to commit to the use of an approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
* Use of any psychotropic medication within four weeks of visit 1, day -14 and throughout the study.
* Use of dietary supplements containing any of the following: lutein, ginkgo biloba, St. John's wort, ginseng, gotu kola (Indian pennywort); daily doses of vitamin E (≥30 mg/d) or folic acid (≥400 ug/d); thiamine, riboflavin, and/or pyridoxine (≥2 mg/d); and eicosapentaenoic acid (EPA), docosahexaenoic acid or a combination of EPA + DHA (≥500 mg/d) within 2 weeks prior to screening.
* Subject has had exposure to any non-registered drug product within 30 days prior to the screening visit and throughout the study.
* Recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >60g (men) / 40g (women) pure alcohol per day (7 / 5.5 units).
* Subject has a known allergy or sensitivity to study product or any ingredients of the study product or meals provided.
* The subject is unable to perform the tests on the COMPASS System during training to the established acceptable levels for participation in this type of study.
* Use of stevia extract sweetened products/drinks or stevia leaves within 1 month of the study

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Associative / Visual Memory (Name to Face Recall (COMPASS)) | Day 0 (baseline) to day 28
  Associative / Visual Memory Task on a computer. Outcome measurements: Change of accuracy and speed of response from baseline measurement to 1 month
Associative / Visual Memory (Name to Face Recall (COMPASS)) | Day 0 (baseline) to day 56
  Associative / Visual Memory Task on a computer. Outcome measurements: Change of accuracy and speed of response from baseline measurement to 2 months
Associative / Visual Memory (Name to Face Recall (COMPASS)) | Day 0 (baseline) to day 77
  Associative / Visual Memory Task on a computer. Outcome measurements: Change of accuracy and speed of response from baseline measurement to 3 months
Visual Memory (Picture Recognition (COMPASS)) | Day 0 (baseline) to day 28
  Visual Memory Tasks on a computer: Outcome measurement: Change in percent correct from baseline measurement to 1 month
Visual Memory (Picture Recognition (COMPASS)) | Day 0 (baseline) to day 56
  Visual Memory Tasks on a computer: Outcome measurement: Change in percent correct from baseline measurement to 2 months
Visual Memory (Picture Recognition (COMPASS)) | Day 0 (baseline) to day 77
  Visual Memory Tasks on a computer: Outcome measurement: Change in percent correct from baseline measurement to 3 months
Working and Spatial Memory ('Sternberg' Numeric Working Memory task (COMPASS)) | Day 0 (baseline) to day 28
  Working and Spatial Memory Tasks on a computer. Outcome measurements: Change of speed and accuracy of performance from baseline measurement to 1 month
Working and Spatial Memory ('Sternberg' Numeric Working Memory task (COMPASS)) | Day 0 (baseline) to day 56
  Working and Spatial Memory Tasks on a computer. Outcome measurements: Change of speed and accuracy of performance from baseline measurement to 2 months
Working and Spatial Memory ('Sternberg' Numeric Working Memory task (COMPASS)) | Day 0 (baseline) to day 77
  Working and Spatial Memory Tasks on a computer. Outcome measurements: Change of speed and accuracy of performance from baseline measurement to 3 months
Working and Spatial Memory ('Corsi Blocks'(COMPASS)) | Day 0 (baseline) to day 28
  Working and Spatial Memory Tasks on a computer. Outcome measurement: Change of span score from baseline measurement to 1 month
Working and Spatial Memory ('Corsi Blocks'(COMPASS)) | Day 0 (baseline) to day 56
  Working and Spatial Memory Tasks on a computer. Outcome measurement: Change of span score from baseline measurement to 2 months
Working and Spatial Memory ('Corsi Blocks'(COMPASS)) | Day 0 (baseline) to day 77
  Working and Spatial Memory Tasks on a computer. Outcome measurement: Change of span score from baseline measurement to 3 months
Executive Function and Verbal Memory (Peg and Ball Task (COMPASS)) | Day 0 (baseline) to day 28
  Executive Function and Verbal Memory Tasks on a computer. Outcome measurements: Change of accuracy, thinking time and speed of performance from baseline measurement to 1 month
Executive Function and Verbal Memory (Peg and Ball Task (COMPASS)) | Day 0 (baseline) to day 56
  Executive Function and Verbal Memory Tasks on a computer. Outcome measurements: Change of accuracy, thinking time and speed of performance from baseline measurement to 2 months
Executive Function and Verbal Memory (Peg and Ball Task (COMPASS)) | Day 0 (baseline) to day 77
  Executive Function and Verbal Memory Tasks on a computer. Outcome measurements: Change of accuracy, thinking time and speed of performance from baseline measurement to 3 months
Executive Function and Verbal Memory (Delayed Word Recognition (COMPASS)) | Day 0 (baseline) to day 28
  Executive Function and Verbal Memory Tasks on a computer. Outcome measurements: Change of accuracy and speed of response from baseline measurement to 1 month
Executive Function and Verbal Memory (Delayed Word Recognition (COMPASS)) | Day 0 (baseline) to day 56
  Executive Function and Verbal Memory Tasks on a computer. Outcome measurements: Change of accuracy and speed of response from baseline measurement to 2 months
Executive Function and Verbal Memory (Delayed Word Recognition (COMPASS)) | Day 0 (baseline) to day 77
  Executive Function and Verbal Memory Tasks on a computer. Outcome measurements: Change of accuracy and speed of response from baseline measurement to 3 months

SECONDARY OUTCOMES:
Attention and Concentration (Choice Reaction Time (COMPASS)) | Day 0 (baseline) to day 28
  Attention and Concentration Tasks on a computer. Outcome measurement:
  Change of speed of response from baseline to 1 month.
Attention and Concentration (Choice Reaction Time (COMPASS)) | Day 0 (baseline) to day 56
  Attention and Concentration Tasks on a computer. Outcome measurement:
  Change of speed of response from baseline to 2 months.
Attention and Concentration (Choice Reaction Time (COMPASS)) | Day 0 (baseline) to day 77
  Attention and Concentration Tasks on a computer. Outcome measurement:
  Change of speed of response from baseline to 3 months.
Attention and Concentration (Rapid Visual Information Processing (COMPASS)) | Day 0 (baseline) to day 28
  Attention and Concentration Tasks on a computer. Outcome measurement:
  Change of accuracy, false alarms, speed of response from baseline to 1 month.
Attention and Concentration (Rapid Visual Information Processing (COMPASS)) | Day 0 (baseline) to day 56
  Attention and Concentration Tasks on a computer. Outcome measurement:
  Change of accuracy, false alarms, speed of response from baseline to 2 months.
Attention and Concentration (Rapid Visual Information Processing (COMPASS)) | Day 0 (baseline) to day 77
  Attention and Concentration Tasks on a computer. Outcome measurement:
  Change of accuracy, false alarms, speed of response from baseline to 3 months.
Bond-Lader Visual Analog Scales (VAS) of Mood | Day 0 (baseline) to day 28
  This questionnaire of 16 analogue scales derives three factors that assess change in self-rated alertness, self-rated calmness and self-rated contentment. (presented within COMPASS) Outcome measurement: Change of these parameters from baseline to 1 month.
Bond-Lader Visual Analog Scales (VAS) of Mood | Day 0 (baseline) to day 56
  This questionnaire of 16 analogue scales derives three factors that assess change in self-rated alertness, self-rated calmness and self-rated contentment. (presented within COMPASS) Outcome measurement: Change of these parameters from baseline to 2 months.
Bond-Lader Visual Analog Scales (VAS) of Mood | Day 0 (baseline) to day 77
  This questionnaire of 16 analogue scales derives three factors that assess change in self-rated alertness, self-rated calmness and self-rated contentment. (presented within COMPASS) Outcome measurement: Change of these parameters from baseline to 3 months.
Profile of Mood States (POMS) Questionnaire | Day 0 (baseline) to day 28
  The POMS provides scales of tension-anxiety, depression-dejection, anger
  -hostility, vigor-activity, fatigue-inertia and confusion-bewilderment. A score will be obtained from each and a single score of "mood disturbance" will be computed. (paper and pencil) Outcome measurement: Change of these parameters from baseline to 1 month.
Profile of Mood States (POMS) Questionnaire | Day 0 (baseline) to day 56
  The POMS provides scales of tension-anxiety, depression-dejection, anger
  -hostility, vigor-activity, fatigue-inertia and confusion-bewilderment. A score will be obtained from each and a single score of "mood disturbance" will be computed. (paper and pencil) Outcome measurement: Change of these parameters from baseline to 2 months.
Profile of Mood States (POMS) Questionnaire | Day 0 (baseline) to day 77
  The POMS provides scales of tension-anxiety, depression-dejection, anger
  -hostility, vigor-activity, fatigue-inertia and confusion-bewilderment. A score will be obtained from each and a single score of "mood disturbance" will be computed. (paper and pencil) Outcome measurement: Change of these parameters from baseline to 3 months.
Prospective and Retrospective Memory Questionnaire (PRMQ) | Day 0 (baseline) to day 28
  Subjects will be asked about their subjective 'prospective' and 'retrospective' memory performance - paper and pencil Outcome measurement: Change of memory scores from baseline to 1 month.
Prospective and Retrospective Memory Questionnaire (PRMQ) | Day 0 (baseline) to day 56
  Subjects will be asked about their subjective 'prospective' and 'retrospective' memory performance - paper and pencil Outcome measurement: Change of memory scores from baseline to 2 months.
Prospective and Retrospective Memory Questionnaire (PRMQ) | Day 0 (baseline) to day 77
  Subjects will be asked about their subjective 'prospective' and 'retrospective' memory performance - paper and pencil Outcome measurement: Change of memory scores from baseline to 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, Prof, Principal Investigator — Director of the 'Brain, Performance and Nutrition Research Centre', Northumbria University, UK; Crystal Haskell, PhD, Principal Investigator — Associate Director of the 'Brain, Performance and Nutrition Research Centre', Northumbria University, UK
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom